CLINICAL TRIAL: NCT04354740
Title: Predictors of Coronary Revascularization Outcomes in Type 2 Diabetic Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rabab Emad Ahmed Mohmed Mashhour, Assistant lecturer of internal medicine, Assiut University
Other Study IDs: coronary revascularization,DM2
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2 With Acute Coronary Syndrom
MeSH Terms: conditions — Diabetes Mellitus | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A : Diabetic: group is subdivided into 2sub-groups: Group 1: Group: underwent PCI(Primary or Rescue) Group 2: underwent CABG Patients diagnosed as multivessel disease or left main coronary artery lesion will be included in the study
  Interventions: Procedure: with percutaneous coronary intervention (PCI) are with new-generation drug-eluting stents (DES)
- Group B: Non diabetic: group is subdivided into 2sub-groups: Group 1: Group: underwent PCI(Primary or Rescue) Group 2: underwent CABG Patients diagnosed as multivessel disease or left main coronary artery lesion will be included in the study
  Interventions: Procedure: with percutaneous coronary intervention (PCI) are with new-generation drug-eluting stents (DES)

INTERVENTIONS:
Procedure: with percutaneous coronary intervention (PCI) are with new-generation drug-eluting stents (DES) — II-PCI:
  -Coronary angiography and intervention will be done according to the European guidelines of ACS revascularization.
  III-CABG:
  Other Names: coronary artery bypass grafting (CABG) with maximal use of arterial grafts

SUMMARY:
* To explore the metabolic outcomes of PCI versus CABG in diabetic patients presented by ACS.
* To verify the diagnostic and prognostic value of speckle tracking echocardiography in early detection of MACE after ACS in diabetic patients treated by 2 modalities.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) doubles the risk of cardiovascular disease and about 75% of deaths in diabetic patients are due to coronary artery disease. Studies performed during the 1980's and 90's demonstrated increasing short and long-term mortality in diabetic patients undergoing CABG compared with non-diabetic patients. However, more recently, reports have shown a significant reduction in mortality among patients with diabetes. Alexander Kogan etal., 2018 Cardiac revascularization in patients with stable coronary artery disease (CAD) is an important therapeutic intervention for the improvement of symptoms and prognosis. Prior to revascularization, patients must receive guideline-recommended medical therapy due to its established benefits. Thomas Nyström etal.,2018 Also notable is that the best current revascularization results achieved with percutaneous coronary intervention (PCI) are with new-generation drug-eluting stents (DES) and for coronary artery bypass grafting (CABG) with maximal use of arterial grafts. The multitude of studies for revascularization comparing PCI and CABG cannot provide a single solution for the entire spectrum of patients with stable CAD. Nevertheless, CABG results in more complete revascularization than PCI, particularly in complex multivessel CAD, which often is observed in patients with diabetes. Thomas Nyström etal., 2018 Approximately 25% of all patients who undergo multivessel revascularization have diabetes. A number of studies have demonstrated that CABG should be the preferred strategy for multivessel revascularization in patients with diabetes. In this group, CABG leads to improved survival rates and a reduced risk of myocardial infarction and repeat revascularization compared with revascularization with PCI. In the BARI (Bypass Angioplasty Revascularization Investigation) trial, a subset of 353 patients with diabetes who underwent PCI had almost a doubled 5-year mortality compared with those who underwent CABG. However, if only saphenous vein grafts were used as conduits, cardiac mortality was similar to that with PCI, demonstrating the importance of arterial grafting. It was further demonstrated in the BARI 2D (Bypass Angioplasty Revascularization Investigation 2 Diabetes) study that among patients with diabetes, prompt revascularization by CABG significantly reduced major CV events compared with intensive medical treatment alone. In contrast, there was no difference in CV events between patients who underwent PCI and patients who received only intensive medical treatment.Thomas Nyström etal.,2018 Pathological left ventricular remodeling (LVR) was the common characteristic of most cardiovascular diseases. It clinically defined as the adverse changes in LV mass, volume, and geometry after myocardial injury, which could be considered to be an adaptive response to cardiac performance inadequacy and a marker of poor prognosis in patients with underlying LV dysfunction. In recent years, the impact of non hemodynamic factors on cardiac structure and function, such as obesity and other metabolic disorder, had been gradually valued. Van Bilsen et al even proposed a theory of "metabolic remodeling." This theory held that glycolipid metabolism disturbance could change the metabolic pathway of myocardial energy and finally lead to LV remodeling and dysfunction. Qingqing Wang etal.,2018 Myocardial strain quantification by speckle tracking echocardiography has been well validated. It is a validated and accurate measure of regional systolic LV function.It has also been shown to be superior to visual assessment of wall motion in detection and quantification of regional systolic function. Strain and other deformation parameters are sensitive tools for detection of ischemia. It is hypothesized that global and regional left ventricular2D strain by speckle tracking echocardiography (STE) facilitates an early and accurate non-invasive tool to predict the presence of acute coronary artery occlusion in patients with non ST-segment elevation myocardial infarction (NSTEMI). Viola William Keddeas,etal 2016

ELIGIBILITY:
Inclusion Criteria:

* This study includes all patients (middle aged according to WHO 55 years of age) presented by ACS (STEMI , Non STEMI) from July 2020 to June2021 in both CCU Of Internal Medicine Departemennt and and EL Orman Assiut University Hospital of Cardiology and Cardiothoracic Surgery.

ACS was defined and patients were managed according to the European Guidelines . Patients with acute chest pain and persistent (>20 min) ST-segment elevation, i.e., STEMI generally reflected an acute total coronary occlusion. All patients received immediate myocardial reperfusion treatment by primary coronary intervention and angioplasty or fibrinolytic therapy, as appropriate. Patients with acute chest pain but no persistent ST-segment elevation, referred to as Non-STEMI included transient ST-segment elevation, persistent or transient ST-segment depression ,T-wave inversion, flat T waves or pseudo-normalized T waves or completely normal ECG at admission. Thygesen, K.; etal.2019

Exclusion Criteria:

* -Ranal disease ie stage 3,4 or on dialysis.
* Advanced hepatic diseases ie(child B,C)
* Poor echo window including morbid obesity.
* Age >18 and more than 55 years old
* Patients with previous history of significant valvular diseases,atrial fibrillation
* EF less than 40%

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: This study includes all patients (middle aged according to WHO 55 years of age) presented by ACS (STEMI , Non STEMI)
  Those patients are divided to:
  Group A : Diabetic Group B: Non diabetic
  Then each group is subdivided into 2sub-groups:
  Group 1: Group: underwent PCI(Primary or Rescue) Group 2: underwent CABG Patients diagnosed as multivessel disease or left main coronary artery lesion will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACEs) | 12 mounths
  Rate of myocardial infarction (MI), Rate of revascularization, Rate of cerebrovascular events"stroke"

SECONDARY OUTCOMES:
In hospital mortality | 12mounths
  Rate of death (mortality rate)after CABG or PCI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel SA, Deepa M, Shivashankar R, Ali MK, Kapoor D, Gupta R, Lall D, Tandon N, Mohan V, Kadir MM, Fatmi Z, Prabhakaran D, Narayan KMV. Comparison of multiple obesity indices for cardiovascular disease risk classification in South Asian adults: The CARRS Study. PLoS One. 2017 Apr 27;12(4):e0174251. doi: 10.1371/journal.pone.0174251. eCollection 2017. PMID 28448582
- [Background] Lu H, Tang B, Zhou Y, Xu C, Bundhun PK, Tang Z, Bao H. Short-Term Versus Long-Term Adverse Cardiovascular Outcomes Post Percutaneous Coronary Intervention in Patients with Insulin-Treated Type 2 Diabetes Mellitus: A Simple Meta-Analysis. Diabetes Ther. 2019 Aug;10(4):1487-1497. doi: 10.1007/s13300-019-0656-9. Epub 2019 Jun 29. PMID 31256352
- See also: (2018) 17:151 Impact of type 2 diabetes mellitus on short- and long-term mortality after coronary artery bypass surgery — https://cardiab.biomedcentral.com/articles/10.1186/s12933-018-0796-7
- See also: 2018. PCI or CABG in Stable Patients With Multivessel CAD and Diabetes — https://www.acc.org/latest-in-cardiology/articles/2018/03/27/08/51/pci-or-cabg-in-stable-patients-with-multivessel-cad-and-diabetes